CLINICAL TRIAL: NCT02739412
Title: Efficacy of Low Dose, Subcutaneous Interleukin-2 (IL-2) to Expand Endogenous Regulatory T-Cells in Liver Transplant Recipients
Brief Title: Efficacy of Low Dose, SubQ Interleukin-2 (IL-2) to Expand Endogenous Regulatory T-Cells in Liver Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Michael Curry, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016P000086
Record Dates: First submitted 2016-04-05; First posted 2016-04-15 (Estimated); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interleukin-2 (Experimental): IL-2 (Interleukin-2; Aldesleukin; Proleukin) administered daily as a single subcutaneous injection 0.30 MIU per meter squared body surface area for a duration of 4 weeks.
  Interventions: Biological: Interleukin-2

INTERVENTIONS:
Biological: Interleukin-2 — Subjects will self-administer low dose IL-2 as subQ injection (0.30 MIU per meter squared body surface area) for 4 weeks.
  Other Names: IL-2; Aldesleukin; Proleukin

SUMMARY:
The purpose of this investigation is to study if very low dose IL-2, given to liver transplant patients by subcutaneous (under the skin) injections, over a 4 week period of time, will cause an increase in the number of Treg cells in the blood.

DETAILED DESCRIPTION:
A common complication of organ transplantation is 'rejection' of the transplanted organ. This occurs when the body's immune system tries to attack (or reject) the transplanted organ.

Drugs known as immunosuppressants (anti-rejection medications) are prescribed for patients after transplantation to prevent rejection. But, anti-rejection medications are associated with significant side effects including high blood pressure, high blood sugars, and high cholesterol - all of which may increase the risk of heart and vascular complications. Anti-rejection medications also increase the long-term risk of some types of cancer.

Sometimes, liver transplant patients who stop taking anti-rejection medications do not experience rejection of their transplanted liver and the liver keeps working. These patients are said to "tolerate" the transplanted liver, and this condition is referred to as "tolerance". Doctors are working to learn more about why some liver transplant patients develop tolerance after receiving a transplant, while others do not.

Studies have shown that patients who develop "tolerance" have an increase in a type of immune cell called regulatory T-cells or "Tregs". This means Tregs may be important in preventing rejection of a transplanted organ.

Studies have also shown that a human cytokine (a type of protein), called interleukin-2 (IL-2) aids in increasing the number of Treg cells in the body, and IL-2 has been given to patients to successfully treat disorders of the immune system such as graft vs host disease - a serious condition sometimes seen in patients after bone marrow transplantation.

The purpose of this investigation is to study if low dose IL-2, given to liver transplant patients by subcutaneous (under the skin) injections, over a 4 week period of time, will cause an increase in the number of Treg cells in the blood.

In addition, investigators will learn about the kinds of side effects low dose IL-2 will cause and how severe those side effects will be.

ELIGIBILITY:
Inclusion criteria:

1. Adult liver transplant recipients 2-4 years post transplantation
2. Male or female adult, age 18 - 65 years
3. Stable dosage of suppressant therapy for 1 month prior to study.

Exclusion criteria:

1. Recipient of multiple transplants (including solid organ, stem-cell, and bone marrow)
2. Serum liver panel (ALT, AST, Alkaline Phosphatase and Total Bilirubin) > 2 x ULN,
3. Serum creatinine > 1.5 x ULN,
4. eGFR of < 40 ml/min,
5. Detectable hepatitis viral load,
6. Abnormal ECG with clinically significant findings per study physician's judgement,
7. Active infection,
8. Presence or history of autoimmunity disorders,
9. Evidence of allograft rejection,
10. Liver biopsy or fibroscan evidence of advanced stage liver fibrosis (> Stage 2 Fibrosis),
11. Presence or history of cardiac or pulmonary disease,
12. Pregnant or nursing (lactating) women,
13. Health condition precludes participation in trial at study physician's judgment,
14. Inability to give consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Curry, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Study Medication Arm: Single arm, prospective, open label efficacy and safety of a 4-weeks course of low dose IL-2 to expand TRegs in liver transplant recipients with stable liver function.
Period: Overall Study
Arm/Group | Active Study Medication Arm
Started | 6
Completed | 5
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: 6 patients were enrolled. 5 patients completed the efficacy analysis, and 6 patients were included in the safety analysis.
Groups:
- Open Label. Active Study Treatment Arm: IL-2 (Interleukin-2; Aldesleukin; Proleukin) administered daily as a single subcutaneous injection 0.30 MIU per meter squared body surface area for a duration of 4 weeks.
Arm/Group | Open Label. Active Study Treatment Arm
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 54 [46 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6
CD3T cells (%PBMC) [Median (Inter-Quartile Range); unit: %PBMC] — Population: 1 patient withdrew from the study after 1 dose due to adverse event and was not included in the efficacy analysis.
  %PBMC
    number analyzed (Participants) | 5
    (all) | 53.74 [51.22 to 61.12]
CD4 T cells (% PBMC) [Median (Inter-Quartile Range); unit: %PBMC] — Population: 1 patient withdrew from the study after 1 dose due to adverse event and was not included in the efficacy analysis.
  %PBMC
    number analyzed (Participants) | 5
    (all) | 25.29 [17.68 to 28.44]
CD8 T cells (%PBMC) [Median (Inter-Quartile Range); unit: %PBMC] — Population: 1 patient withdrew from the study after 1 dose due to adverse event and was not included in the efficacy analysis.
  %PBMC
    number analyzed (Participants) | 5
    (all) | 28.05 [21.94 to 32.78]
CD19 B cells (%PBMC) [Median (Inter-Quartile Range); unit: %PBMC] — Population: 1 patient withdrew from the study after 1 dose due to adverse event and was not included in the efficacy analysis.
  %PBMC
    number analyzed (Participants) | 5
    (all) | 4.84 [3.93 to 9.17]
CD56 NK (%PBMC) [Median (Inter-Quartile Range); unit: %PBMC] — Population: 1 patient withdrew from the study after 1 dose due to adverse event and was not included in the efficacy analysis.
  %PBMC
    number analyzed (Participants) | 5
    (all) | 6.37 [5.26 to 16.91]
Monocyte/Dendritic cells (% PBMC) [Median (Inter-Quartile Range); unit: %PBMC] — Population: 1 patient withdrew from the study after 1 dose due to adverse event and was not included in the efficacy analysis.
  %PBMC
    number analyzed (Participants) | 5
    (all) | 12.82 [10.78 to 18.19]
NKT (%PBMC) [Mean (Inter-Quartile Range); unit: %PBMC] — Population: 1 patient withdrew from the study after 1 dose due to adverse event and was not included in the efficacy analysis.
  %PBMC
    number analyzed (Participants) | 5
    (all) | 13.56 [3.41 to 17.01]
CD4Treg (% of PBMC) [Median (Inter-Quartile Range); unit: %PBMC] — Peripheral blood lymphocytes % of CD4 Tregs Population: 1 patient withdrew from the study after 1 dose due to adverse event and was not included in the efficacy analysis.
  %PBMC
    number analyzed (Participants) | 5
    (all) | 0.44 [0.275 to 0.75]
CD4 conventional T cells (% of CD4 cells) [Median (Inter-Quartile Range); unit: %PBMC] — Population: 1 patient withdrew from the study after 1 dose due to adverse event and was not included in the efficacy analysis.
  %PBMC
    number analyzed (Participants) | 5
    (all) | 97.34 [96.31 to 98.80]
CD4 Treg cells (% CD4 T cells) [Median (Inter-Quartile Range); unit: %PBMC] — Population: 1 patient withdrew from the study after 1 dose due to adverse event and was not included in the efficacy analysis.
  %PBMC
    number analyzed (Participants) | 5
    (all) | 2.13 [1.04 to 3.12]
Alanine aminotransferase (ALT) [Mean (Full Range); unit: units of ALT/L] — Normal range is 0-40 U/L. Above 40U/L is abnormal.
  units of ALT/L | 19 [15 to 22]
White Blood Cell count (WBC) [Median (Inter-Quartile Range); unit: cells *10^9/L] | 5.85 [5.1 to 5.9]
Platelet count [Median (Inter-Quartile Range); unit: platelets /uL] | 162,000 [113,000 to 195,000]
Hematocrit [Median (Inter-Quartile Range); unit: %] | 39 [38.1 to 39.7]
Time from transplant [Median (Full Range); unit: years] | 2.85 [2.09 to 3.47]

OUTCOME MEASURES:

1. Primary Outcome: Regulatory T-Cell Count
Description: Peripheral Blood Mononuclear Cell Flow Cytometry
Time Frame: baseline, week 2, week 4, week8, week12
Population: The efficacy analysis was performed on 5 patients. 1 patient withdrew from the study due to an adverse event before any efficacy data was obtained.6 patients were enrolled, 66% male with a median age of 54 years. Median time from transplant was 2.8 years. Five patients were on tacrolimus monotherapy and 1 patients was on tacrolimus and mycophenolate mofetil.
Measure: Median (Inter-Quartile Range); unit: percentage of PBMC
Groups:
- Open Label. Active Study Treatment Arm: All patients received IL-2
Arm/Group | Open Label. Active Study Treatment Arm
Number analyzed (Participants) | 5
percentage of PBMC
  Baseline CD4Tred (%PBMC) | 0.44 [0.27 to 0.75]
  Wk2 CD4Treg (%PBMC) | 3.71 [2.95 to 4.48]
  Wk4 CD4Treg (%PBMC) | 3.57 [2.53 to 3.59]
  Wk8 CD4Treg (%PBMC) | 0.6 [0.42 to 1.37]
  Wk12 CD4Treg (%PBMC) | 0.64 [0.44 to 1.28]
Statistical Analysis 1: Comparison: Open Label. Active Study Treatment Arm; This is an open label feasibility study to assess the efficacy and safety of a 4 week course of daily subcutaneous IL-2 injections to increase peripheral blood CD4 Tregs. Results are expressed as median, IQR and comparison were performed using one way or two-way ANOVA, followed by Tukey's multiple comparison test. For all comparisons, a p< 0.05 was considered significant; Test type: Superiority — Power calculations were not performed in this study; p < 0.01, ANOVA

2. Primary Outcome: % Increase in CD4 Tregs
Description: % CD4 T Regs were measured at several time points after IL-2 administration.
Time Frame: baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of CD4 T cells
Arm/Group | Active Study Medication Arm
Number analyzed (Participants) | 5
percentage of CD4 T cells
  Baseline CD4Treg (%CD4Tcells) | 2.13 [1.04 to 3.12]
  Wk2 CD4Treg (%CD4Tcells) | 13.15 [11.53 to 19.02]
  Wk4 CD4Treg (%CD4Tcells) | 11.93 [8.88 to 15.94]
  Wk8 CD4Treg(%CD4Tcells) | 2.79 [1.51 to 5.18]
  Wk12 CD4Treg (%CD4Tcells) | 2.63 [1.75 to 4.94]

3. Secondary Outcome: Differential Immune Cell Count
Description: Peripheral Blood Mononuclear Cell Flow Cytometry
Time Frame: baseline, 2 weeks, 4 weeks, 8 weeks, 12 Weeks
Measure: Median (Inter-Quartile Range); unit: percentage of PMBC
Arm/Group | Active Study Medication Arm
Number analyzed (Participants) | 5
percentage of PMBC
  Baseline CD3Tcells (%PBMC) | 53.74 [51.22 to 61.12]
  Wk2 CD3Tcells (%PBMC) | 57.05 [43.29 to 64.80]
  Wk4 CD3Tcells (%PBMC) | 53.69 [47.02 to 58.79]
  Wk8 CD3Tcells (%PBMC) | 58.00 [49.32 to 61.33]
  Wk12 CD3 Tcells (%PBMC) | 53.35 [47.08 to 63.17]
  Baseline CD4Tcells (%PBMC) | 25.59 [17.68 to 28.44]
  Wk2 CD4Tcells (%PBMC) | 23.7 [16.06 to 29.94]
  Wk4 CD4Tcells (%PBMC) | 26.11 [17.61 to 30.02]
  Wk8 CD4Tcells (%PBMC) | 26.91 [17.86 to 31.73]
  Wk12 CD4Tcells (%PBMC) | 26.08 [17.43 to 33.03]
  Baseline CD8Tcells (%PBMC) | 28.05 [21.94 to 32.78]
  Wk2 CD8Tcells (%PBMC) | 22.9 [18.46 to 29.94]
  Wk4 CD8Tcells (%PBMC) | 22.9 [18.26 to 24.57]
  Wk8 CD8Tcells (%PBMC) | 24.88 [22.23 to 29.51]
  Wk12 CD8Tcells (%PBMC) | 23.23 [20.34 to 29.00]
  Baseline CD19Bcells (%PBMC) | 4.84 [3.93 to 9.175]
  Wk2 CD19Bcells (%PBMC) | 4.84 [4.35 to 7.70]
  Wk4 CD19Bcells (%PBMC) | 3.63 [3.54 to 9.00]
  Wk8 CD19Bcells (%PBMC) | 6.16 [4.73 to 11.65]
  Wk12 CD19Bcells (%PBMC) | 6.63 [4.41 to 12.40]
  Baseline CD56NKcells (%PBMC) | 6.37 [5.26 to 16.91]
  Wk2 CD56NKcells (%PBMC) | 12.53 [8.58 to 19.51]
  Wk4 CD56NKcells (%PBMC) | 11.72 [9.71 to 18.91]
  Wk8 CD56NKcells (%PBMC) | 6.95 [4.68 to 16.62]
  Wk12 CD56NKcells (%PBMC) | 6.09 [4.86 to 18.72]
  Baseline NKTcells (%PBMC) | 13.56 [3.41 to 17.01]
  Wk2 NKTcells (%PBMC) | 11.75 [2.94 to 12.88]
  Wk4 NKTcells (%PBMC) | 9.33 [3.40 to 12.42]
  Wk8 NKTcells (%PBMC) | 10.69 [3.12 to 12.21]
  Wk12 NKTcells (%PBMC) | 11.58 [2.95 to 12.04]
  Baseline Monocytes/Dendritic | 12.82 [10.78 to 18.19]
  Wk2 Monocytes/Dendritic cells (%PBMC) | 9.00 [6.17 to 23.54]
  Wk4 Monocytes/Dendritic (%PBMC) | 12.87 [9.25 to 21.35]
  Wk8 Monocytes/Dendritic (%PBMC) | 11.77 [10.60 to 21.05]
  Wk12 Monocytes/Dendritic (%PBMC) | 12.35 [10.09 to 22.83]

4. Other Pre Specified Outcome: Kidney Function Serum Panel (> 1.5 x Upper Limit Normal)
Description: Number of participants with a serum creatinine > 1.5 x upper limit of normal through week 36
Time Frame: 2 weeks, 4 weeks, 8 weeks, 12 weeks, 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Interleukin-2
Number analyzed (Participants) | 6
Participants
  Week 2 | 1
  week 4 | 0
  week 8 | 0
  week 12 | 0
  week 36 | 0

5. Other Pre Specified Outcome: Liver Function Serum Panel (> 2 x Upper Limit Normal)
Description: Number of patients with a serum amino alaninetransferase > 2 x upper limit of normal through week 36
Time Frame: week 2, 4 week, week 8, week12, week36
Measure: Count of Participants; unit: Participants
Arm/Group | Active Study Medication Arm
Number analyzed (Participants) | 6
Participants
  week 2 | 0
  week 4 | 0
  week 8 | 0
  weeks 12 | 0
  week 36 | 0

ADVERSE EVENTS:
Time Frame: 36 weeks
Description: Adverse events and serious adverse events were collected at day 1, 3, week 1, 2, 3, 4, 8, 12 and 36
Arm/Group | Active Study Medication Arm
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Study Medication Arm (N=6)
Legionella disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Study Medication Arm (N=6)
arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Injection site reaction (Skin and subcutaneous tissue disorders) | 6 (6)
Fatigue (General disorders) | 2 (2)
eosinophilia (Blood and lymphatic system disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Mouth Ulcer (Gastrointestinal disorders) | 1 (1)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1)
Fracture radius (Musculoskeletal and connective tissue disorders) | 1 (1)
abnormal EKG (Cardiac disorders) | 1 (1)
Edema (General disorders) | 1 (1)
Ankle Injury (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The analysis for phenotypic T cell exhaustion was not performed due to inadequate remaining peripheral blood mononuclear cells on all study participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-07): https://cdn.clinicaltrials.gov/large-docs/12/NCT02739412/Prot_SAP_000.pdf
  • Informed Consent Form: date change (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/12/NCT02739412/ICF_001.pdf